CLINICAL TRIAL: NCT05458765
Title: A Phase II Acceptability Study of Oral Emtricitabine/Tenofovir Alafenamide (F/TAF) vs Emtricitabine/Tenofovir Disoproxil Fumarate (F/TDF) for the Prevention of HIV Acquisition in Adolescent Girls and Young Women (AGYW)
Brief Title: Project Engage: Oral PrEP Acceptability
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: CONRAD (Other); FHI 360 (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CONRAD B20-151
Record Dates: First submitted 2022-06-10; First posted 2022-07-14 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2023-08

CONDITIONS: Acceptability of Health Care; Adherence, Medication
Keywords: PrEP; HIV
MeSH Terms: conditions — Patient Acceptance of Health Care; Medication Adherence | interventions — emtricitabine tenofovir alafenamide; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Complete blinding is not possible, however, to the extent possible, clinicians or study staff who collect adverse event data will be blinded to the randomization assignments to limit bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- F/TAF (Active Comparator): daily oral tablet
  Interventions: Drug: emtricitabine/tenofovir alafenamide
- F/TDF (Active Comparator): daily oral tablet
  Interventions: Drug: Emtricitabine / Tenofovir Disoproxil Oral Tablet

INTERVENTIONS:
Drug: emtricitabine/tenofovir alafenamide — 200mg/25mg tablet, once daily dosing for 24 weeks
  Other Names: Descovy
  Arms: F/TAF
Drug: Emtricitabine / Tenofovir Disoproxil Oral Tablet — 200mg/300mg tablet, once daily dosing for 24 weeks
  Other Names: Truvada
  Arms: F/TDF

SUMMARY:
This study is a two-arm open label acceptability study that will examine acceptability of, and adherence to, once daily dosing regimen of F/TDF (Truvada) and an investigational once daily dosing regimen of F/TAF (Descovy) under standard of care counselling. The study will recruit approximately 330 healthy, HIV negative, AGYW in up to three sites in Africa. Eligible participants will be randomized 1:1 to receive F/TAF 200 mg/25 mg or F/TDF 200 mg/300 mg for once daily oral administration for 24 weeks.

Study visits will take place according to standard of care at month 1, month 3 and month 6. Acceptability and adherence will be assessed by questionnaires and DBS at months 3 and 6; questionnaires will assess acceptability of product attributes; perceived pill side effects; ease of pill-taking and reasons for missed pills, and future interest in PrEP use beyond the trial context. Exit interviews at the final visit and additional qualitative interviews and focus group discussions with a subset of participants as well as other key stakeholders will further inform potential differences in acceptability and adherence between the two products. Data collection will also focus on gathering insights and input from participants that will aid uptake and continuation and inform future programming of oral PrEP.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age 15 to 24 years (inclusive)
2. Literate, per local standards, to English and/or local language
3. In general good health, per participant reported medical history and investigator judgement, without any clinically significant systemic disease including but not limited to: significant liver disease or hepatitis, gastrointestinal disease, kidney disease, osteoporosis or bone disease (e.g., pathologic bone fractures not related to trauma), autoimmune disorder, and diabetes.
4. Willing to give voluntary informed consent and sign an informed consent form
5. Sexually active or considered at risk of acquiring HIV
6. Willing and able to comply with protocol requirements, including swallowing tablets
7. Total body weight >35 kg
8. eGFR or Creatinine Clearance of >60 mL/min according to the Cockcroft-Gault formula
9. Has not used oral PrEP ever (PrEP naïve) or in the past 6 months
10. If pregnant, must be considered a healthy, singleton pregnancy, considered low risk by local standard of obstetric practices

Exclusion Criteria:

1. Positive test for HIV or HBsAg
2. Signs or symptoms of acute HIV infection
3. Use of ARV PrEP within the past 180 days
4. History of sensitivity or allergy to any component of the study drug products
5. Systemic use in the last two (2) weeks or anticipated use during the course of the study of any restricted products
6. Known current drug or alcohol abuse which could impact study compliance
7. Grade 2 or higher laboratory abnormality, except for CrCl 60-90 mL/min, per the Division of AIDS, National Institute of Allergy and Infectious Disease (DAIDS) Table for Grading the Severity of Adverse Events, or clinically significant laboratory abnormality as determined by the clinician or study PI
8. Abnormal finding on laboratory or physical examination or a social or medical condition in the volunteer, which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data
9. Participation in any other investigational trial with use of a drug/device within the last 30 days or planned participation in any other investigational trial with use of a drug/device during the study
10. History of pathological bone fracture
11. Pregnant <33 weeks gestation; breastfeeding with infant >6 months old
12. Has a sexual partner confirmed to be HIV positive per participant report

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 330 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Compare the discontinuation rate between arms | 3 months
  Acceptability will be assessed by discontinuation of study product

SECONDARY OUTCOMES:
Adherence to study product | 3 months
  Concentrations of TFV-DP and FTC-TP in dried blood spots (DBS)

OTHER OUTCOMES:
Psychometric scales predictive validity of adherence to study product | 3 and 6 months
  Participant classifications based on correlations between screening scales and DBS drug concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Doncel, MD,PhD, Study Director — CONRAD/EVMS; Homaira Hanif, PhD, Principal Investigator — CONRAD/EVMS
Locations (3):
- South Africa (2):
  - MatCH Research Unit, Durban, KwaZulu-Natal
  - CAPRISA Vulindlela, Pietermaritzburg, KwaZulu-Natal
- Harare Health and Research Consortium (HHRC), Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No